CLINICAL TRIAL: NCT05942768
Title: Efficacy and Safety of Anti-PD-1 Antibody Plus Regorafenib in Refractory Microsatellite Stable Metastatic Colorectal Cancer: a Retrospective Single-arm Cohort Study
Brief Title: Anti-PD-1 Antibody Plus Regorafenib in Refractory Microsatellite Stable Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REGOPD-1-Hunan
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: Colorectal cancer;regorafenib;anti-PD-1 antibodies
MeSH Terms: interventions — regorafenib; Programmed Cell Death 1 Receptor; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: regorafenib plus anti-PD-1 antibodies — The patients were treated orally with regorafenib (80 mg once daily for 21 days on/7 days off, over a 28-day cycle), combined with 1 of the 5 anti-PD-1 antibodies (i.e., nivolumab, pembrolizumab, camrelizumab, sintilimab, or toripalimab). The anti-PD-1 antibody was administered intravenously on day 1, and its recommended dosage was as follows: nivolumab: 240 mg, every 2 weeks; pembrolizumab, camrelizumab, and sintilimab: 200 mg every 3 weeks; and toripalimab: 240 mg every 3 weeks
  Other Names: programmed cell death protein 1; immune checkpoint inhibitor

SUMMARY:
Managements for refractory proficient mismatch repair (pMMR) or microsatellite stable (MSS) metastatic colorectal cancer (mCRC) were still challenging and controversial. Our study sought to investigate the efficacy and safety of anti-PD-1 antibodies plus regorafenib in refractory pMMR/MSS mCRC between July 2019 and June 2021 at the Hunan Cancer Hospital.

DETAILED DESCRIPTION:
We retrospectively analyzed the efficacy and safety of 103 pMMR/MSS mCRC patients treated with at least one dose of anti-PD-1 antibodies plus regorafenib (80 mg once daily for 21 days on/7 days off 28 days as a cycle) between July 2019 and June 2021 at the Hunan Cancer Hospital. All patients had previously received at least second-line treatment. The patients were evaluated by computed tomography every 2 or 3 treatment cycles until progression or being lost to follow-up. The primary end point was overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* 1.Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded).

  2. Have progressed from at least 2 lines of standard treatment,including fluoropyrimidines, irinotecan, oxaliplatin, with or without targeted drugs, like bevacizumab and cetuximab (only for RAS wild-type).

  3.Has measurable or non-measurable disease as defined by RECIST version 1.1 4.Is able to swallow oral tablets. 5.Estimated life expectancy ≥12 weeks. 6.Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1 7. Has adequate organ function.

Exclusion Criteria:

* 1.Pregnancy, lactating female or possibility of becoming pregnant during the study.

  2.Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy (excluding alopecia, and skin pigmentation).

  3.Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.

  4.Has severe or uncontrolled active acute or chronic infection. 5.Known carriers of HIV antibodies. 6.Confirmed uncontrolled arterial hypertension or uncontrolled or symptomatic arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population were the patients treated with at least 1 cycle of anti-PD-1 antibodies plus regorafenib between July 2019 and June 2021 at the Hunan Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of commencement of treatment and the date of death due to any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the date of commencement of treatment and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.
Overall response rate (ORR) | Approximately 12 months
  Overall response rate (ORR) was regarded as the proportion of complete responses (CRs) and partial responses (PRs) according to RECIST version 1.1 criteria and using investigator's tumor assessment
Disease control rate (DCR) | Approximately 12 months
  Disease control rate has been defined as the addition of (CR + PR) rate and also stable disease (SD) rate
Treatment-Related Adverse Events (TRAE) | Approximately 12 months
  Treatment-Related Adverse Events (TRAE) as assessed by CTCAE v5.0, including serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for principal investigator or correspondence author]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author.